CLINICAL TRIAL: NCT05370638
Title: Discharge in the AM: A Randomized Controlled Trial of Physician Rounding Styles to Improve Hospital Throughput and Length of Stay
Brief Title: Discharge in the AM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Denver Health and Hospital Authority (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 19-1607
Record Dates: First submitted 2022-04-25; First posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Hospitalism; Flow or Discharge
Keywords: hospitalist; patient flow; early discharge; discharge before noon; inpatient

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rounding on discharging patients first (Experimental): Rounding on discharging patients meant that the attending physician and accompanying team (i.e. if they were working with advanced practice providers or learners) would prioritize seeing any patients that were going to discharge that day.
  Interventions: Other: Rounding on discharging patients first
- usual practice (No Intervention): Usual practice was categorized as: seeing discharging patients first, sickest patients, decompensating patients, new patients (i.e. patients admitted to their team overnight), or based on geography.

INTERVENTIONS:
Other: Rounding on discharging patients first — Rounding on discharging patients meant that the attending physician and accompanying team (i.e. if they were working with advanced practice providers or learners) would prioritize seeing any patients that were going to discharge that day. The attending could break protocol if needed for patient care purposes and this was tracked each day.
  Arms: rounding on discharging patients first

SUMMARY:
As hospitals around the country continue to work to manage a high patient census, provider prioritization of discharges is one low cost mechanism to help improve patient throughput and patient length of stay. The investigators conducted a prospective randomized study to understand if this commonly utilized approach to expedite care results in earlier discharges and lower hospital lengths of stay while also understanding the impact on other patient care (such as test and consult order times on other patients that the physician is caring for).

DETAILED DESCRIPTION:
Hospitals around the country face bottlenecks and capacity issues. When hospitals are successful at managing high capacity this allows for increased access for patients who need this higher level of care and expertise.

Unfortunately, hospital discharges frequently occur in the afternoon or evening hours and can adversely affect patient flow throughout the hospital which, in turn, can result in delays in care, medication errors, increased mortality, longer lengths of stay, higher costs, lower patient satisfaction, and decreased access to care at these facilities. While some of the delays in discharges result, appropriately, from the caring of other patients and conducting the necessary tasks and assessments for acutely ill patients, previous work also identified that providers may be able to prioritize their work in a different way in order to facilitate this throughput. The investigators aim to conduct a randomized controlled trial of physician rounding style at three institutions in order to: (1) determine if prioritizing discharging patients first will result in earlier discharges and decreased lengths of stay, (2) determine if prioritizing discharges first will cause other care delays or affect patient experience and, (3) determine factors that contribute to physician ability to prioritizing discharges first. The study is a prospective, multi-center, cluster randomized trial designed to test the effects of rounding on discharging patients first compared to usual practice and will utilize an effectiveness-implementation hybrid approach. The investigators will recruit hospitalist attending physicians from three hospitals in the US to be randomized to one of two rounding styles: (1) prioritize discharges first and (2) usual practice. The main outcome measure will be discharge order time. Secondary outcomes will be length of stay and lab/diagnostic test order time. Additionally, the investigators will study how team composition (teaching, non-teaching, teams with advanced practice providers), team census (i.e. the number of patients a provider is caring for), and number of admissions affect the ability for providers to prioritize discharges first.

Through qualitative methods the investigators will also gain an understanding from physicians as to why or why not they were able to prioritize discharges first. This study will add to the evidence to either support or negate the practice of prioritizing discharges. There have been no randomized studies to date that have addressed these issues. Additionally, the investigators aim to understand how team composition and census affect discharge times. Institutions across the country will be able to utilize these findings to help refine current rounding models. The investigators believe these findings will be pivotal for clinicians to be more willing to change their practice style. The investigators also believe this study will aid in the understanding of what factors may function as facilitators and barriers of earlier discharges.

ELIGIBILITY:
Inclusion Criteria:

Physicians:

-Hospital Medicine attending-level physicians who consented to participate and patients

Patients:

* At least 18 years of age
* Admitted to a Medicine service and assigned by standard practice to a general medical hospitalist team including a provider who agreed to participate in the study

Exclusion Criteria:

-Patients assigned, by standard practice, to a general medical hospitalist team and on the team of providers who chose not to participate in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Physician discharge order time | From the midnight of the day the patient was discharged until time the patient had a discharge order placed, assessed up to 6 months from the start of the study.
  Physician discharge order time entered into the electronic health record

SECONDARY OUTCOMES:
Patient discharge time | From the midnight of the day the patient was discharged until the time the patient was discharged from the hospital, assessed up to 6 months from the start of the study.
  The time the patient left their hospital bed/actually discharged from care in the hospital
Patient length of stay | From the time that the patient was admitted to hospital until time the patient had a discharge order placed, assessed up to 6 months from the start of the study.
  The total length of stay in hours
Average time of day of orders for imaging, consults, or procedures were entered by participating physicians into the electronic health record | From the midnight of the day each day to the time of day each patient had an order placed for imaging, consults, or procedures, assessed up to 6 months from the start of the study.
  average time of day over the course of each patient's hospitalization that orders for imaging, consults, or procedures were entered by participating physicians

CONTACTS AND LOCATIONS:
Overall Officials: Marisha Burden, MD, Principal Investigator — University of Colorado School of Medicine
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Burden M, Gundareddy VP, Kauffman R, Keach JW, McBeth L, Raffel KE, Rice JD, Washburn C, Kisuule F, Keniston A. Assessing the impact of workload and clinician experience on patient throughput: A multicenter study. J Hosp Med. 2025 May;20(5):471-478. doi: 10.1002/jhm.13555. Epub 2024 Nov 26. PMID 39588662